CLINICAL TRIAL: NCT03553199
Title: Pilot Study on a New Endoscopic Platform for the ESD of Colorectal Lesions: Tissue Retraction System
Brief Title: Study on a New Endoscopic Platform for the ESD of Colorectal Lesions: Tissue Retraction System
Acronym: TRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRS
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Tissue Retraction System
Keywords: Tissue Retraction System; Colorectal polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- TRS (Experimental): TRS, Tissue resection system
  Interventions: Device: TRS, Tissue Retraction System

INTERVENTIONS:
Device: TRS, Tissue Retraction System — Tissue Retraction System

SUMMARY:
Endoscopic submucosal dissection (ESD) is an endoscopic technique that allows the removal of lesions of the gastrointestinal tract. The European Society of Gastrointestinal Endoscopy (ESGE) suggests to consider ESD for the removal of colorectal lesions that cannot be removed enbloc with standard polypectomy or endoscopic mucosal resection (EMR) and for lesions that are > 20 mm in diameter, with a high probability of having a limited submucosal invasion.

ESD is a technically difficult and time-consuming procedure that is very difficult to learn and to perform, but it allows higher enbloc resection rates compared to other endoscopic techniques and is less invasive than surgery requiring less length of hospital stay.

Recently, several new techniques and devices have been developed to facilitate ESD and to overcome difficulties related to challenging situations. The main difficulties are related to the instability of the operating field, due to the physiologic peristalsis, and to the loss of traction, due to the single operating channel.

DETAILED DESCRIPTION:
Tissue Retraction System (TRS, Boston scientific) is a new endoscopic platform, that consists of an expandable and dynamically-controlled intra-luminal chamber, mounted on a flexible overtube, and two associated specifically designed retractor graspers. The system is front-loaded over the colonoscope and introduced into the colon. When the target area is reached, the retractor system is deployed creating an expanded, optimally reconfigured and stable operating field around the target lesion. Then endoscopic removal of the lesion is performed using available endoscopic instruments (injection needles, knives, snares, etc) through the operating channel of the colonoscope with assistance of two retractor graspers. Each accessory within the TRS can be moved forward and backward, left or right, rotated 360 degrees, and can be advanced out and pulled in, regardless of the TRS.

The investigators hypothesize that the TRS can improve visualization of lesions and stabilize the work environment by allowing retraction and tissue resection during ESD.

TRS is a new device not yet commercially available, thus no study has been already performed in humans to evaluate its feasibility and safety to speed up the ESD of left colon and rectum lesions.

The investigator's proposal is to perform a pilot study to evaluate the feasibility, the efficacy and the safety in patients undergoing ESD of colorectal lesions with the assistance of the TRS.

ELIGIBILITY:
Inclusion Criteria:

* left colon and rectal lesions matching the criteria of ESD removal: depressed/flat elevated morphology and irregular or nongranular surface pattern, larger than 20 mm; lesions that cannot be optimally and radically removed with standard polypectomy or EMR
* age ≥18 years
* ability to sign the informed consent

Exclusion Criteria:

* deep submucosal invasion diagnosed by distorted pit (Kudo's type V) and/or capillary (Sano's type III) patterns [5];
* poor general condition (American Society of Anesthesiologists score ≥ 3);
* coagulation disorders;
* pregnancy and breastfeeding;
* inability to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is the feasibility, defined as the technical success rate, to perform an enbloc ESD with the assistance of the TRS. | 9 months

SECONDARY OUTCOMES:
Secondary endpoints are: the efficacy, defined as the rate of lesions removed enbloc and the rate of curative ESD (with an R0 resection); the safety, defined as the rate of adverse events (AEs). | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Italy

IPD SHARING:
Plan to Share IPD: No